CLINICAL TRIAL: NCT03699436
Title: Effectiveness of an Intervention Program With Electric Stimulation Therapy in Patients With Raynaud's Phenomenon: a Randomized Clinical Trial
Brief Title: Effectiveness of Electric Stimulation Therapy in Raynaud's Phenomenon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Encarnación Aguilar Ferrandiz, Research and teaching staff of the University of Granada, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ray-2016
Record Dates: First submitted 2018-10-04; First posted 2018-10-09 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Raynaud Phenomenon; Raynaud Disease
Keywords: Vascular alterations; Galvanic current; Pain; Peripheral blow flow; Temperature; Upper limb functionality; Central Sensitization; Pain catastrophizing.; Number of attacks
MeSH Terms: conditions — Raynaud Disease; Pain | interventions — Electric Stimulation Therapy; Control Groups

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Electric Stimulation Therapy Group (Experimental): The experimental group will receive an electrotherapy treatment with galvanic current in their hands. Electrotherapy with galvanic current has vasodilator action.
  Interventions: Other: Electrotherapy with Galvanic Current
- Control Group (Active Comparator): The control group will be subjected to a conservative treatment. These patients will continue to take their usual medication and will not receive electrotherapy treatment
  Interventions: Other: Control without Electric Stimulation Therapy

INTERVENTIONS:
Other: Electrotherapy with Galvanic Current — The experimental group will receive an electrotherapy treatment with galvanic current in their hands.This protocol will be administered at weekly sessions of 30 minutes with a period of 3 times / week with a total of 20 sessions, distributed over a 7-week period. They will be evaluated at baseline, after the end of the last treatment session and after two months of follow-up.
  Other Names: Electric Stimulation Therapy
  Arms: Electric Stimulation Therapy Group
Other: Control without Electric Stimulation Therapy — The control group continue with their usual conservative and pharmacological treatment and will not receive electrotherapy treatment. They will be evaluated too at baseline, after the end of the last treatment session and after two months of follow-up.
  Other Names: Control Group
  Arms: Control Group

SUMMARY:
The purpose of this study is to analyze the effects of an intervention with galvanic electrical current on the number of attacks , temperature, pain, peripheral blow flow and upper limb functionality in patients with Raynaud's Phenomenon in comparison to a control group that will maintain their habitual treatment.

DETAILED DESCRIPTION:
Raynaud's Phenomenon is a disorder that causes pain and functional limitation in people who suffer it.

Investigators considerer that the application of an electrotherapy intervention with galvanic current, thanks to its vasodilator action, will produce clinically significant improvements in the number of attacks, temperature and blood flow of patients with Raynaud's Phenomenon, which can lead to a decrease in pain associated, frequency and severity of ischemic attacks and therefore an improvement in the functionality of the upper limbs.

The experimental group will receive an electrotherapy treatment using galvanic current. To apply the treatment, we will place the patient seated, with their hands inside two containers filled with water up to the limit of their nails without touching them. Next we will connect the electrodes and apply a galvanic current for 10 minutes, there will be a minute of rest for the patient while we change the polarity of this current and we will apply it another 10 minutes. The intensity of the current depends on the threshold of the patient.

The control group will maintain their usual conservative and pharmacological treatment without receiving electrotherapy

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years of age.
* Being diagnosed with Primary or Secondary Raynaud Phenomenon according to the criteria established by LeRoy-Medsger.
* A history of at least one year of regular attacks of pallor or acral cyanosis caused by exposure to cold and/or stress.
* Having signed the informed consent document and willingness to participate in the study

Exclusion Criteria:

* Presence of skin alterations such as stings, scars, ulcers or gangrene in the examined area.
* Suffering upper limb entrapment syndrome, central nervous system polyneuropathy, Hypothyroidism, renal failure, cerebral or cardiac ischemic disease.
* History of drug or alcohol abuse.
* Pregnant or breastfeeding women.
* Use of vibratory tools.
* Participants with tumour process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Number of Raynaud´s Phenomenon attacks | Seven Weeks
  Change from baseline at the Number of Raynaud´s Phenomenon attacks

SECONDARY OUTCOMES:
Temperature in the affected areas in patients with Raynaud´s Disease | Seven weeks
  Change from baseline temperature in the infrared thermography in patients with Raynaud´s Disease
Temperature in the affected areas in patients with Raynaud´s Disease | Fifteen weeks
  Change from baseline temperature in the infrared thermography in patients with Raynaud´s Disease
Temperature in the Cold Stress Test | Seven weeks
  Change from temperature in the Cold Stress Test
Temperature in the Cold Stress Test | Fifteen weeks
  Change from temperature in the Cold Stress Test
Pain Intensity: Visual Analog Scale | Seven weeks
  Change from baseline in pain in the Visual Analog Scale. Score range between 0-10 cm where 0 is in considerer no pain and 10 is the worst pain imaginable.
Pain Intensity: Visual Analog Scale | Fifteen weeks
  Change from baseline in pain in the Visual Analog Scale. Score range between 0-10 cm where 0 is in considerer no pain and 10 is the worst pain imaginable.
Central Sensitization | Seven weeks
  Change from baseline in the Central Sensitization Inventory. The cumulative score ranges from 0 to 100.Higher scores indicate increased frequency and severity of the symptoms.
Central Sensitization | Fifteen weeks
  Change from baseline in the Central Sensitization Inventory. The cumulative score ranges from 0 to 100.Higher scores indicate increased frequency and severity of the symptoms.
Pain Catastrophizing | Seven weeks
  Change from baseline in the Pain Catastrophizing Scale. Score range is from 0 to 52; higher scores indicate a greater frequency of catastrophic thoughts.
Pain Catastrophizing | Fifteen weeks
  Change from baseline in the Pain Catastrophizing Scale. Score range is from 0 to 52; higher scores indicate a greater frequency of catastrophic thoughts.
Oxygen Saturation | Seven weeks
  Change from baseline in Oxygen Saturation
Oxygen Saturation | Fifteen weeks
  Change from baseline in Oxygen Saturation
Arterial blood flow | Seven weeks
  Change from baseline in Arterial blood flow in the radial and ulnar artery
Arterial blood flow | Fifteen weeks
  Change from baseline in Arterial blood flow in the radial and ulnar artery
Upper limb disability | Seven Weeks
  Change from baseline in the Disabilities of the Arm, Shoulder and Hand Questionnaire. The score ranges from 0 (no disability) to 100 (most severe disability). Higher scores indicate a greater level of disability and severity.
Upper limb disability | Fifteen Weeks
  Change from baseline in the Disabilities of the Arm, Shoulder and Hand Questionnaire. The score ranges from 0 (no disability) to 100 (most severe disability). Higher scores indicate a greater level of disability and severity.

CONTACTS AND LOCATIONS:
Overall Officials: Mª Encarnacion ME Aguilar Ferrandiz, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- University of Granada, Granada, Spain